CLINICAL TRIAL: NCT07156578
Title: A Long-Term, Open-Label Extension Study of Bivamelagon in Participants With Hypothalamic Obesity (HO)
Brief Title: A Long-Term Study of Bivamelagon in Participants With Hypothalamic Obesity (HO)
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-MC72-002
Record Dates: First submitted 2025-08-25; First posted 2025-09-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hypothalamic Obesity
MeSH Terms: conditions — Sexual Infantilism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bivamelagon (open-label) (Experimental)
  Interventions: Drug: Bivamelagon

INTERVENTIONS:
Drug: Bivamelagon — daily dose of oral bivamelagon

SUMMARY:
This is a long-term, open-label extension study of bivamelagon in participants with Hypothalamic Obesity (HO) who have transitioned from the index study, LG-MCCL005. The study will last up to 2 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Completed LG-MCCL005 and participant demonstrated adequate safety and tolerability in that study as determined by the Investigator.
* Agree to use a highly effective form of contraception and follow contraception requirements throughout the study and for 90 days after.

Key Exclusion Criteria:

* Willing to remain off of: CYP3A4 inhibitors, strong CYP3A4 inducers, and P-glycoprotein inhibitors or substrates for the duration of the study.
* In the opinion of the Investigator, participant is not suitable to participate in the study.

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2028-04-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of bivamelagon as assessed by the number and frequency of AEs | Baseline to up to 2 years

SECONDARY OUTCOMES:
Mean change and mean percentage change from Baseline in BMI in participants ≥18 years of age. | Baseline to up to 2 years
Mean change in BMI z-score in participants >18 years of age. | Baseline to up to 2 years
Mean change in and mean percentage change in weight | Baseline to up to 2 years
Mean change in percentage of the 95th percentile of BMI in participants <18 years of age. | Baseline to up to 2 years
Percentage of patients who achieve ≥5%,≥10%, ≥15%, and ≥20% reduction in BMI from baseline | Baseline to up to 2 years
Mean change from Baseline in Physical function (and total score) for the Impact of Weight on Quality of Life-Lite (IWQoL) in participants ≥18 years of age | Baseline to up to 2 years
Change from Baseline in total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, and triglycerides | Baseline to up 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (9):
- United States (6):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Columbia University, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- United Kingdom (3):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - University of Cambridge, Cambridge
  - Great Ormond Street Hospital for Children, London

IPD SHARING:
Plan to Share IPD: No